CLINICAL TRIAL: NCT06714266
Title: A Prospective, Single-arm, Phase II Clinical Trial to Evaluate the Efficacy and Safety of Trilaciclib in Preventing Hematopoietic Suppression in Patients with Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma Receiving Either Single Chemotherapy or Chemotherapy Combined with Immunotherapy/targeted Therapy.
Brief Title: Trilaciclib in Preventing Hematopoietic Suppression in Patients with Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Man Hu, Chief Physician/Professor, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SDZLEC2024-264-02
Record Dates: First submitted 2024-11-20; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC)
Keywords: Head and neck squamous cell carcinoma; Chemotherapy induced myelosuppression; Trilaciclib
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — trilaciclib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients were treated with Trilaciclib + chemotherapy ± immune/targeted therapy (Experimental): Trilaciclib 240mg/m2, intravenous infusion for 30 minutes, completed within 4 hours before daily chemotherapy; Chemotherapy regimen: FP regimen (cisplatin/carboplatin +5-FU regimen: cisplatin 75mg/m2 D1, D2, D3 or carboplatin AUC 5, intravenous infusion D1; 5-FU 1000 mg/m2, intravenous infusion, D1-4; Q3W); TP regimen (cisplatin/carboplatin +5-FU regimen: cisplatin 75mg/m2 D1, D2, D3 or carboplatin AUC 5, intravenous infusion D1; Docetaxel 75mg/m2 or albumin paclitaxel 200mg, IV infusion, D1, 8; Q3W). The specific dose can be adjusted according to the situation.
  Immunotherapy: pembrolizumab 200mg q2w Targeted therapy: cetuximab (400mg/m2 qw 250mg/m2 qw) Some patients could be treated with maintenance therapy, and the treatment regimen was immunotherapy or targeted therapy combined with treaclib.
  Interventions: Drug: Trilaciclib

INTERVENTIONS:
Drug: Trilaciclib — Trilaciclib 240mg/m2, intravenous infusion for 30 minutes, completed within 4 hours before daily chemotherapy; Chemotherapy regimen: FP regimen (cisplatin/carboplatin +5-FU regimen: cisplatin 75mg/m2 D1, D2, D3 or carboplatin AUC 5, intravenous infusion D1; 5-FU 1000 mg/m2, intravenous infusion, D1-4; Q3W); TP regimen (cisplatin/carboplatin +5-FU regimen: cisplatin 75mg/m2 D1, D2, D3 or carboplatin AUC 5, intravenous infusion D1; Docetaxel 75mg/m2 or albumin paclitaxel 200mg, IV infusion, D1, 8; Q3W). The specific dose can be adjusted according to the situation.
  Immunotherapy: Pembrolizumab 200mg q2w Targeted therapy: cetuximab (400mg/m2 qw 250mg/m2 qw) Some patients can be treated with maintenance therapy, and the treatment regimen is immunotherapy or targeted therapy combined with Trilaciclib
  Other Names: chemotherapy; immune/targeted therapy

SUMMARY:
This prospective, single-arm, exploratory, phase II study was designed to evaluate the efficacy and safety of Trilaciclib in reducing chemotherapy-induced neutropenia in patients with recurrent or metastatic head and neck squamous cell carcinoma. Eligible subjects screened by the inclusion and exclusion criteria will receive chemotherapy alone or combined with immune/targeted therapy and Trilaciclib for 4-6 cycles of continuous treatment. If the efficacy is not progressive after 4-6 cycles of treatment, the investigators can combine with Trilaciclib during immune and/or targeted maintenance therapy according to the specific conditions of the subjects until disease progression or intolerance. The efficacy of Trilaciclib will be evaluated by the incidence of grade ≥3 neutropenia during chemotherapy as the primary endpoint.

After the progression of treatment, if the subjects were treated with chemotherapy for subsequent treatment and were considered to be able to use Trilaciclib according to the evaluation of the investigator, the use of treaclib could be considered until the subjects had disease progression again or were intolerant to treatment.

DETAILED DESCRIPTION:
Head and neck squamous cell carcinoma (HNSCC) is the seventh most common malignant tumor in the world, accounting for 5% of all head and neck cancers in China. Among them, head and neck squamous cell carcinoma accounts for 90% of all head and neck malignant tumors, including nasopharyngeal carcinoma, oropharyngeal cancer, hypopharyngeal cancer, lip cancer, laryngeal cancer, nasal cavity cancer, paranasal sinus cancer, etc. Due to the complex anatomical and physiological structure of the head and neck, head and neck squamous cell carcinoma (HNSCC) is a highly heterogeneous group of malignant tumors. In all head and neck squamous cell carcinoma, more than 60% of patients are initially diagnosed as locally advanced (stage Ⅲ-Ⅳ, excluding M1). After comprehensive treatment, 40%-60% of patients will eventually develop local recurrence or distant metastasis, and the 5-year survival rate is less than 50%. Platinum-based chemotherapy remains the main treatment option. The first-line treatment is immune/targeted combination chemotherapy.

Chemotherapy induced myelosuppression (CIM) is a common and important side effect in cancer treatment. 80% of chemotherapy drugs can cause bone marrow suppression, infection, bleeding, fatigue and other side effects, which seriously reduce the quality of life of patients, increase the economic burden, and may also lead to the reduction or delay of chemotherapy, which directly affects the anti-tumor efficacy of chemotherapy. In a retrospective analysis of patients with small-cell lung cancer, non-Hodgkin's lymphoma, head and neck cancer, and breast cancer by Yanli Li et al., 77.5% of patients had a high risk for Febrile neutropenia (FN) during chemotherapy. 18.8% of patients were hospitalized due to infection during the first course of treatment. For each additional day of continuous chemotherapy, the risk of hospitalization due to infection increased by 28% in patients with CIN 3/4, respectively, and the risk was 30% in patients with CIN 4. A study of 1111 patients with early-stage breast cancer treated with adjuvant chemotherapy from 13 large administrative, academic, and community practice centers showed that 61.2% of patients had delayed and reduced doses of chemotherapy due to: Neutropenia, 60.7% of patients with delayed chemotherapy and dose reduction caused by neutropenia will have neutropenia again, which seriously affects the survival and prognosis of patients.

CIM is mainly reflected in erythropenia, neutropenia and thrombocytopenia, and the existing prevention methods for chemotherapy-induced bone marrow suppression have limitations. Recombinant human granulocyte coloby stimulating fator (G-CSF) can prevent febrile neutropenia, but may increase the risk of adverse reactions such as musculoskeletal pain. rhTPO and rhIL-11 can prevent chemotherapy-induced thrombocytopenia, but the operation is complicated and the adverse reactions are serious, especially cardiac toxicity and edema. Currently, there is no effective prevention for erythropenia. In the past, the traditional treatment for bone marrow suppression is not true bone marrow protection. G-CSF is also given after chemotherapy to stimulate the proliferation of surviving progenitor cells, and may even cause the exhaustion of bone marrow hematopoietic reserve function. Dose reduction and delayed administration of chemotherapy drugs are also common clinical measures to cope with CIM. These dose adjustments limit the relative dose intensity of the planned treatment and may reduce the potential benefit of patients. Safe, effective and easy to operate preventive drugs for myelosuppression, especially for thrombocytopenia and anemia, are currently unmet clinical needs.

Trilaciclib is a highly potent, selective, and reversible CDK4/6 inhibitor that protects bone marrow by protecting hematopoietic stem/progenitor cells and lymphocytes during systemic chemotherapy. The proliferation and differentiation of progenitor cells are very dependent on the activity of CDK4/6. When they are exposed to appropriate doses of traC, they will be arrested in the G1 phase of the cell cycle. Therefore, intravenous administration of traC before chemotherapy can protect blood cells from cell cycle-toxic chemotherapy drugs. At the same time, treaclib can protect/enhance the immune system, make lymphocytes temporarily arrest, reduce the apoptosis of T lymphocytes and directly enhance the immune response. Changing the proliferation kinetics and composition of T cell subsets in the tumor is beneficial to enhance the effector function and improve the tumor microenvironment.

This prospective, single-arm, exploratory, phase II study was designed to evaluate the efficacy and safety of Trilaciclib in reducing chemotherapy-induced neutropenia in patients with recurrent or metastatic head and neck squamous cell carcinoma. Eligible subjects screened by the inclusion and exclusion criteria will receive chemotherapy alone or combined with immune/targeted therapy and Trilaciclib for 4-6 cycles of continuous treatment. If the efficacy is not progressive after 4-6 cycles of treatment, the investigators can combine with Trilaciclib during immune and/or targeted maintenance therapy according to the specific conditions of the subjects until disease progression or intolerance. The efficacy of Trilaciclib will be evaluated by the incidence of grade ≥3 neutropenia during chemotherapy as the primary endpoint.After the progression of treatment, if the subjects were treated with chemotherapy for subsequent treatment and were considered to be able to use Trilaciclib according to the evaluation of the investigator, the use of treaclib could be considered until the subjects had disease progression again or were intolerant to treatment.

The research unit of this clinical study is Shandong Cancer Hospital Affiliated to Shandong First Medical University, and it plans to enroll 30 patients with head and neck squamous cell carcinoma. This study protocol has been reviewed and approved by the ethics committee of Shandong Cancer Hospital Affiliated to Shandong First Medical University.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written informed consent was obtained before enrollment.
* 2. Age ≥18 years old, both male and female;
* 3. Recurrent or metastatic head and neck squamous cell carcinoma without prior systemic therapy;
* 4. the presence of at least one measurable lesion;
* 5. ECOG PS = 0-1;
* 6. Expected survival time ≥ 3 months
* 7. Laboratory tests meet the following standards: Hemoglobin ≥ 100 g/L (female), 110g/L (male) Neutrophil count ≥ 2×109/L Platelet count ≥100×109/L; Creatinine ≤ 15mg/L or creatinine clearance (CrCl) ≥ 60 mL/min (Cockcroft-Gault formula); Total bilirubin ≤ 1.5× upper limit of normal value (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN or ≤5× ULN (in patients with liver metastases); Albumin ≥ 30 g/L;
* 8. Women: all women of childbearing potential must have a negative serum pregnancy test during the screening period and must be using a reliable contraceptive method from the time of informed consent until 3 months after the last dose;

Exclusion Criteria:

* 1. Patients with known allergies to any of the drugs in the study;
* 2. Participated in other drug clinical trials within 4 weeks before the study;
* 3. a history of major bleeding, with any bleeding event of CTCAE4.0 grade 3 or above within 4 weeks before screening;
* 4. patients with hypertension that is not well controlled by single antihypertensive medication (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg); 8. Clinically significant (e.g., active) cardiovascular disease - e.g., cerebrovascular accident (≤ 6 months before randomization), myocardial infarction (≤ 6 months before randomization), unstable angina, congestive heart failure of New York Heart Association (NYHA) class II or higher, or severe arrhythmias that could not be controlled with medications or that could potentially affect trial treatment;
* 5. Previous arterial/venous thrombosis events occurred within 6 months before screening, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis (except venous thrombosis caused by intravenous catheterization due to previous chemotherapy, which was judged by the investigator to be cured), and pulmonary embolism;
* 6. Renal insufficiency: urine routine proteinuria > 2+ and confirmed 24-hour urinary protein quantitation > 1.0 g;
* 7. Symptomatic brain metastases (proven or suspected);
* 8. Presence of severe or uncontrolled infection;
* 9. Those who have a history of psychotropic drug abuse and cannot be abstinent or have a history of mental disorder;
* 10. A history of immunodeficiency, including testing positive for HIV, other acquired or congenital immunodeficiency disorders, or a history of organ transplantation; He had a history of autoimmune diseases.
* 11. Use of high-dose glucocorticoids for 4 weeks.
* 12. Patients with previous or current objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severe impairment of pulmonary function, etc.;
* 13. Concomitant medical conditions that, in the investigator's judgment, seriously compromise patient safety or interfere with patient completion of the study. He had received a previous hematopoietic stem-cell or bone marrow transplant
* 14. Allergy to the study drug or its components;
* 15. Those who were deemed unsuitable for the study by the investigator.
* 16. Electrolyte disorder, low calcium, low potassium, low phosphorus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Grade ≥3 neutropenia during chemotherapy alone or combined with immune/targeted therapy | 2year

SECONDARY OUTCOMES:
The incidence of grade 4 neutropenia during treatment | 2year
Objective response rate (ORR) | 2year
The incidence of adverse events | 2year
  Safety and tolerability

IPD SHARING:
Plan to Share IPD: No